CLINICAL TRIAL: NCT06251622
Title: Comparison of Muscle Function and Physical Activity Levels Between People With Cystic Fibrosis and Healthy Individuals in the Modern Era of CFTR (Cystic Fibrosis Transmembrane Conductance Regulator) Modulators: A Case-Control Study
Brief Title: Muscle Function and Physical Activity in the Modern Era of Cystic Fibrosis
Acronym: MUCOMUSCLE
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_1226
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; CFTR modulators; Physical activity; Muscle function
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with Cystic fibrosis treated with CFTR modulators: Children (over 10 years old) and adults with cystic fibrosis, with a stable clinical condition and no contraindications to engaging in moderate-intensity physical activities (PA).
  Interventions: Other: Volumetric ultrasound of the quadriceps and fitting of an accelerometer
- Healthy individuals: Healthy children (over 10 years old) and adults without known diseases (chronic respiratory, cardiovascular, metabolic, renal, or neuromuscular diseases) that may affect their peripheral muscle strength.

INTERVENTIONS:
Other: Volumetric ultrasound of the quadriceps and fitting of an accelerometer — The research procedure will simply involve a volumetric ultrasound of the quadriceps and the fitting of an accelerometer (watch worn on the wrist) for one week (collection of usual physical activities).
  Groups: People with Cystic fibrosis treated with CFTR modulators

SUMMARY:
Cystic fibrosis (CF) is characterized by various extrapulmonary manifestations, including altered skeletal muscle function, with both quantitative (e.g. reduced muscle mass) and qualitative (e.g. impaired oxidative function) impairments that may have a negative impact on exercise tolerance and quality of life. These abnormalities have traditionally been related to disease (e.g. systemic inflammation) or behavioral factors (e.g. increased physical inactivity). However, most of the studies that observed these abnormalities and tried to shed light on the underlying factors were either small or conducted before the widespread of CFTR (Cystic fibrosis transmembrane conductance regulator) modulators that have profound impact on the trajectory of the disease. While several studies suggested that the major recent improvements in therapeutics, including highly effective CFTR modulators, may have positive effects on skeletal muscle function, either directly (e.g. improved mitochondrial function) or indirectly (e.g. reduction in physical inactivity), no studies to date have thoroughly investigated this issue in a representative sample of people with CF. The absence of recent data on muscle function and physical activity levels casts doubt on the relevance of recommendations on exercise training in this population that were published before the widespread use of highly effective CFTR modulators. This study aims to compare muscle function, measured according to the latest recommendations of the European Cystic Fibrosis Society (Saynor et al., 2023), and physical activity of children and adults with CF under CFTR modulators, compared to age- and sex-matched healthy individuals. We hypothesize that the strength, endurance, muscle power, and physical activity levels of individuals with cystic fibrosis, treated with CFTR modulators, remain reduced compared to healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for inclusion of CF patients:

  * Diagnosis of cystic fibrosis
  * Treated with CFTR modulator therapy
  * Men and women (children or adults) aged 10 years or older
  * Affiliated with or entitled to social security coverage
  * For people ≥ 18 years old: participant expressing its oral non-opposition
  * For minor child (<18 years old): participant and its legal representative expressing their oral non-opposition
* Criteria for inclusion of healthy subjects:

  * Men and women (children or adults) aged 10 years or older
  * Affiliated with or entitled to social security coverage
  * For people ≥ 18 years old: participant expressing its oral non-opposition
  * For minor child (<18 years old): participant and its legal representative expressing their oral non-opposition

Exclusion Criteria:

* Exclusion criteria for CF patients:

  * Lack of a stable clinical condition (defined here as the presence of a pulmonary exacerbation and/or a significant change in treatments in the three weeks preceding inclusion in the study).
  * Medical contraindication to engage in moderate-intensity physical activity.
  * Knee joint pain incompatible with the measurement of quadriceps strength.
  * Pregnancy.
* Exclusion criteria for healthy subjects:

  * Known chronic respiratory, cardiovascular, metabolic, renal, or neuromuscular diseases.
  * Presence of benign illnesses and/or acute infections requiring a doctor's visit and occasional treatment in the three weeks preceding inclusion in the study.
  * Medical contraindication to engage in moderate-intensity physical activity.
  * Knee joint pain incompatible with the measurement of quadriceps strength.
  * Pregnancy.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population of patients with cystic fibrosis is selected from the patient cohort at Renée Sabran Hospital, a specialized center for the monitoring and treatment of patients with cystic fibrosis. The healthy individuals will be recruited in the general population from University and Hospital staff (including their children).
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of isometric quadriceps strength (expressed in Newton), performed at René Sabran Hospital (as part of routine clinical practice for people with CF) | Day 0
  The quadriceps strength will be measured on an isometric chair according to the last recommendations of the European Cystic Fibrosis Society (Saynor et al., 2023). Briefly, participants will perform at least three maximal voluntary contractions of the knee extensors, each lasting 4-6s, with a minimal recovery of 1-min between each attempt, with the aim to obtain three maximal quadriceps strength values varying less than 5% (that is usually obtained in less than 6 trials). The highest strength value among these three attempts will be kept for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- HCL - Hôpital Renée Sabran, Hyères, France

IPD SHARING:
Plan to Share IPD: No